CLINICAL TRIAL: NCT00572286
Title: Evaluation of Non-invasive Methods for the Detection of Acute Rejection in Heart Transplant Patients: Use of Echocardiography and Magnetocardiography (MCG) -Pilot Study
Brief Title: Non-invasive Evaluation of Heart Transplant Rejection- Pilot Study
Status: Withdrawn | Type: Observational
Why Stopped: sponsor funding
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: CardioMag Imaging (Industry)
Responsible Party: Kirsten Tolstrup, MD, Cedars-Sinai Medical Center
Other Study IDs: 8144
Record Dates: First submitted 2007-12-12; First posted 2007-12-13 (Estimated); Last update posted 2009-11-17 (Estimated); Status verified 2009-11

CONDITIONS: Advanced Heart Failure; Heart Transplantation
Keywords: heart transplant; advanced heart failure; orthotropic heart transplantation; (MCG) magnetocardiograph; echocardiogram

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: heart transplant patient ( pre or post)

SUMMARY:
The purpose of this research study is to apply new non-invasive, no-risk techniques to a cardiac transplant population for assessment of their reliability in detecting heart transplant rejection.

Graft rejection remains a major factor limiting long-term survival despite continued advancement in the use of immunosuppression. Aggressive surveillance for the detection of acute rejection is therefore necessary. Repeated endomyocardial biopsy (EMB) (at least 11 times the first year after transplantation) remains the only reliable surveillance method available. EMB is expensive, invasive, inconvenient to the patient, and associated with a significant incidence of serious complications. Therefore, it would be very important for patient care if new no-risk methods would prove to be effective in surveillance of rejection.

This research study is designed to measure non-invasive ways to assess rejection along with the standard planned endomyocardial biopsies you will have after heart transplantation. First, the investigators plan to test the effectiveness of the investigational use of the CMI 2406 Magnetocardiograph that has been approved by the U.S Food and Drug Administration (FDA). While the device used in the study is FDA-approved for the non-invasive measurements and recordings of the heart's magnetic field reflecting the heart's electrical currents, it is not yet approved for the specific use of detection of transplant rejection.

DETAILED DESCRIPTION:
Objectives:

The objectives of this study are to test the hypotheses that:

1. Tissue Doppler Imaging, Real time 3D segmental volume measurements, Magnetocardiographic Imaging plus serum markers and T-cell response change when transplant rejection occurs.
2. Tissue Doppler Imaging, Real time 3D segmental volume measurements, Magnetocardiographic Imaging plus serum markers and T-cell response remain stable when no rejection occurs

Background:

General:

Heart transplantation is an advantageous procedure for selected patients with end-stage heart failure. All patients remain on lifetime calcineurin immunosuppressive medications such as cyclosporine or tacrolimus to prevent rejection and extend graft function. Currently, the common practice in managing these patients has been titration of immunosuppressive medications to establish trough levels and clinical response. However, despite the diligent efforts to balance "adequate" immunosuppressive levels with prevention of end-organ toxicity or opportunistic infection; patients still experience acute rejection.

Graft rejection remains a major factor limiting long-term survival despite continued advancement in the use of immunosuppression. Aggressive surveillance using the gold standard of endomyocardial biopsy (EMB) for the detection of acute rejection is therefore necessary. Repeated EMB (a minimum of 11 times the first year after heart transplantation) remains the only reliable surveillance method available. EMB is expensive, invasive, inconvenient to the patient, and associated with a significant incidence of serious complications.

Hyperacute rejection occurs rarely since screening of recipient for anti-donor antibodies has been introduced. However, the focal or diffuse acute cellular rejection is more common and is diagnosed by EMB. The degree or severity of rejections is graded on a scale from 0 to 4 with a grade 3 or more being considered severe. Most acute cellular rejections occur within the first year after transplant. Chronic rejection or allograft arteriopathy occurs later and is monitored by coronary angiography.

Echocardiogram:

Echocardiograms are routinely performed in transplant patients. The findings of increased wall thickness decreased isovolumetric relaxation time and decreased compliance as well as decreased right ventricular (RV) or left ventricular (LV) ejection fraction may indicate rejection, and these parameters may normalize when the rejection resolves.

Tissue Doppler imaging (TDI) measurements are relatively new Doppler techniques for assessing left ventricular diastolic function. Selective measurements of tissue contraction and relaxation velocities at the mitral annulus can detect left ventricular dysfunction more accurately than conventional echocardiography. As left ventricular diastolic dysfunction is an early event during allograft rejection, these techniques may be useful for detecting rejection non-invasively. Few studies have shown that Doppler tissue imaging of the mitral annulus is useful in diagnosing heart transplant rejection (1-3).

Real time 3-dimensional (3D) echocardiography (RT-3D) may be a useful tool in evaluation of patients with coronary artery disease, left ventricular apical thrombi, valvular disease, in guiding intracardiac catheter placement and mitral valvuloplasty. RT-3D, which has recently become widely available, provides dynamic pyramidal data structures that encompass the entire heart and allows four-dimensional assessment of cardiac anatomy and function. It has been shown that this technique is very precise in determination of LV volume, mass and EF measurement and is well correlating with MRI (4-6). Mild changes in LV volume, LV mass and function occur during acute cardiac rejection. This very sensitive technique for assessment of regional volumetric changes has not yet been used for heart transplants monitoring.

Magnetocardiogram:

The Magnetocardiograph (MCG) is a novel imaging modality that may provide a sensitive and objective means to assess alterations in the heart tissue. Because the acute inflammatory process of rejection deleteriously affects myocyte structure and function, we hypothesize that either or both the de- and re-polarization changes will occur in the cardiac cycle with subsequent changes in the cardiac magnetic fields and may give altered readings in the affected patient over time.

Magnetocardiography (MCG) is a new modality which utilizes superconducting quantum interference devices for the detection of the weak magnetic fields (picoTesla range) generated by the heart's electrical currents. The magnetic field map picture, which is created by the measurements of the magnetic field, reflects the electrophysiological state of the heart. When there is an abnormality in cardiac depolarization or repolarization, such as in ischemia or myocarditis, this is reflected in an abnormality in the magnetic field map (7). Although MCG and ECG both measure the cardiac depolarization and repolarization patterns, they have fundamental differences. MCG is most sensitive to tangential currents whereas ECG is most sensitive to radial currents in relation to the chest surface (7-10). Cardiac abnormalities, which interfere with the normal activation and deactivation sequence, such as may occur in acute rejection, increase the contribution of tangential currents. In addition, the MCG detects the vortex currents which are not evident by ECG. Finally, the MCG is less affected by conductivity variations caused by lungs, skin, and muscles and there is no skin electrode contact problem since the device does not come in direct contact with the skin. Therefore, the MCG may be able to detect differences in depolarization and repolarization in a different manner and with a higher sensitivity than the ECG. We speculate that the variation in the magnetic field pattern is due to early subtle changes in cellular mechanisms or metabolism. These changes create a heterogeneous repolarization pattern probably caused by local currents appearing at the border zones between normal and diseased myocardium. This implies that changes in the MCG may appear even earlier in the cascade of rejection than wall motion abnormalities, ECG changes, or changes in serum markers such as troponin.

Schmitz et al reported a sensitivity of 91% and a specificity of 93% for the detection of acute rejection episodes in 15 transplant patients (11). Another study, utilizing a different analysis method, found a sensitivity and specificity of 83% and 84%, respectively for the diagnosis of graft rejection in 12 patients and 6 controls (12).

ELIGIBILITY:
Inclusion Criteria:

* Patients who will have heart transplantation or who have had heart transplantation AND who are scheduled for surveillance biopsies

Exclusion Criteria:

* Patients with Pacemakers or Implantable Cardioverter-Defibrillators(ICD)
* Patients with poor echocardiographic images
* Patients with irregular atrial fibrillation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who will have heart transplantation or who have had heart transplantation
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2005-10; Primary Completion 2009-12 (Estimated); Study Completion 2009-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten Tolstrup, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

REFERENCES:
- [Background] Stengel SM, Allemann Y, Zimmerli M, Lipp E, Kucher N, Mohacsi P, Seiler C. Doppler tissue imaging for assessing left ventricular diastolic dysfunction in heart transplant rejection. Heart. 2001 Oct;86(4):432-7. doi: 10.1136/heart.86.4.432. PMID 11559685
- [Background] Derumeaux G, Douillet R, Redonnet M, Mouton-Schleifer D, Soyer R, Cribier A, Letac B. [Detection of acute rejection of heart transplantation by Doppler color imaging]. Arch Mal Coeur Vaiss. 1998 Oct;91(10):1255-62. French. PMID 9833090
- [Background] Mankad S, Murali S, Kormos RL, Mandarino WA, Gorcsan J 3rd. Evaluation of the potential role of color-coded tissue Doppler echocardiography in the detection of allograft rejection in heart transplant recipients. Am Heart J. 1999 Oct;138(4 Pt 1):721-30. doi: 10.1016/s0002-8703(99)70188-2. PMID 10502219
- [Background] Bu L, Munns S, Zhang H, Disterhoft M, Dixon M, Stolpen A, Sonka M, Scholz TD, Mahoney LT, Ge S. Rapid full volume data acquisition by real-time 3-dimensional echocardiography for assessment of left ventricular indexes in children: a validation study compared with magnetic resonance imaging. J Am Soc Echocardiogr. 2005 Apr;18(4):299-305. doi: 10.1016/j.echo.2004.11.002. PMID 15846155
- [Background] Mannaerts HF, van der Heide JA, Kamp O, Stoel MG, Twisk J, Visser CA. Early identification of left ventricular remodelling after myocardial infarction, assessed by transthoracic 3D echocardiography. Eur Heart J. 2004 Apr;25(8):680-7. doi: 10.1016/j.ehj.2004.02.030. PMID 15084373
- [Background] Kuhl HP, Schreckenberg M, Rulands D, Katoh M, Schafer W, Schummers G, Bucker A, Hanrath P, Franke A. High-resolution transthoracic real-time three-dimensional echocardiography: quantitation of cardiac volumes and function using semi-automatic border detection and comparison with cardiac magnetic resonance imaging. J Am Coll Cardiol. 2004 Jun 2;43(11):2083-90. doi: 10.1016/j.jacc.2004.01.037. PMID 15172417
- [Background] 7.Stroink G, Moshage W, Achenbach S. Cardiomagnetism. In: Andrä W, Nowak H, editors. Magnetism in Medicine.WILEY-VCH Verlag Berlin GmbH. 1998:136-189.
- [Background] Plonsey R. Comparative capabilities of electrocardiography and magnetocardiography. Am J Cardiol. 1972 May;29(5):735-6. doi: 10.1016/0002-9149(72)90179-8. No abstract available. PMID 5021505
- [Background] 9.Hänninen H, Takala P, Mäkijärvi M, et al. Detection of exercise-induced myocardial ischemia by multichannel magnetocardiography in single vessel coronary artery disease. A.N.E. 2000;5:147-157.
- [Background] Hanninen H, Takala P, Korhonen P, Oikarinen L, Makijarvi M, Nenonen J, Katila T, Toivonen L. Features of ST segment and T-wave in exercise-induced myocardial ischemia evaluated with multichannel magnetocardiography. Ann Med. 2002;34(2):120-9. doi: 10.1080/07853890252953518. PMID 12108575
- [Background] 11.Schmitz L, Koch H, Brockmeier K, Müller J, Schüler S, Warnecke H, et al. Magnetocardiographic diagnosis of graft rejection after heart transplantation. In Biomagnetism: Clinical Aspects. Elsevier Science Publishers, Amsterdam. 1992.
- [Background] 12.Achenbach S, Moshage W, Fürst S, Killmann R, Mundl H, Permanetter B et al. Investigation of magnetocardiographic parameters for the detection of graft rejection after heart transplantation. In Biomagnetism: Fundemental research and clinical applications. IOS Press, Amsterdam. 1995.